CLINICAL TRIAL: NCT06080152
Title: Effect of Walker vs Wheeled Device on Mobility After Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Derek Amanatullah, Associate Professor of Orthopaedic Surgery, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 70192
Record Dates: First submitted 2023-07-10; First posted 2023-10-12 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Total Knee Arthroplasty

STUDY DESIGN:
Intervention Model Description: Patient who is using a walker is randomized into two groups:
  1. 12 patients get an A-linker 3 months before surgery (knee arthroplasty)
  2. 12 patients use a walker 3 months before surgery (knee arthroplasty)
  All 24 patients will undergo a total knee Arthroplasty surgery.
  Questionnaires at:
  0 week from randomization into two groups 6 weeks 12 weeks (surgery) 18 weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1 (Experimental): 1. 12 patients get an A-linker 3 months before surgery (knee arthroplasty)
  Interventions: Device: Mobility Tool
- 2 (No Intervention): 2. 12 patients use a walker 3 months before surgery (knee arthroplasty)

INTERVENTIONS:
Device: Mobility Tool — An A-Linker device will be given to 12 patients 3 months before their total knee arthroplasty
  Arms: 1

SUMMARY:
Maneuverability is currently under appreciated by patients who are seeking mobility. This pilot study is examining how patients maneuverability and mobility will change with this novel mobility tool - A-Linker compared to the standard of care walker.

DETAILED DESCRIPTION:
Patients who are using a walker is randomized into two groups:

1. 12 patients get an A-linker 3 months before surgery (knee arthroplasty)
2. 12 patients use a walker 3 months before surgery (knee arthroplasty)

All 24 patients will undergo a total knee Arthroplasty surgery.

Questionnaires at:

0 week from randomization into two groups 6 weeks 12 weeks (surgery) 18 weeks

ELIGIBILITY:
Inclusion Criteria:

* Receiving total knee arthroplasty

Exclusion Criteria:

* Not receiving total knee arthroplasty

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Mobility after surgery | 6 months
  Mobility will be assess using MyPhD linked wearable device. The software will help us capture-
  Steps: # of steps per hour
  Walking/Running distance: per hour

SECONDARY OUTCOMES:
Questionnaire Results | 6 months
  Mobility will be assess using MyPhD linked wearable device. The software will help us capture-
  Steps: # of steps per hour
  Walking/Running distance: per hour
Determining intensity of pain | 6 months
  We plan to use VAS pain scale as measurement scale ( range; 0-10, higher scores correspond to greater pain
Change in knee society score | 6 months
  To assess the effectiveness of the device by calculating Initial knee society score (KSS) and Knee society score at 2 weeks, 3 months and 2 years after surgery. The scale ranges from 0-100 with grading as Score 80-100 - Excellent Score 70-79 - Good Score 60-69 - Fair Score below 60 - Poor
surgery cancellation | 6 months
  To determine if surgery was cancelled as a result of effectiveness of device
Timed up & Go | 6 months
  Calculating Timed up & Go at 6 months visit
Use of gait aide | 6 months
  To assess the effectiveness of the device by examining Gait Aide use at discharge, 2 weeks, 3 months and 2 years after surgery. This is done to examine performance . The gait aide use provident ranges as Nothing > Cane > crutch > walker
Time with Device | 6 months
  Determining compliance of device usage

CONTACTS AND LOCATIONS:
Locations (1):
- 450 Broadway, Redwood City, California, United States